CLINICAL TRIAL: NCT00694148
Title: NT 201 is a Botulinum Toxin Type A Preparation Free of Complexing Proteins. Injected Into the Muscle, NT 201 Causes a Reversible Local Relaxation of the Injected Muscle. Botulinum Toxin Type A is Widely Used for Aesthetic Treatment of Mimic Wrinkles. This Study Will Investigate the Safety and Efficacy of NT 201 in the Treatment of Glabellar Frown Lines.
Brief Title: Safety and Efficacy of NT 201, Free of Complexing Proteins, in the Treatment of Glabellar Frown Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 60201 GL_3001; 2008-000549-73 (EudraCT Number)
Record Dates: First submitted 2008-06-02; First posted 2008-06-10 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Healthy
Keywords: Treatment of glabellar frown lines
MeSH Terms: interventions — incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NT 201 — A Botulinum neurotoxin type A, free of complexing proteins
  Detailed described in study protocol

SUMMARY:
NT 201 is a Botulinum toxin type A preparation free of complexing proteins. Injected into the muscle, NT 201 causes a reversible local relaxation of the injected muscle. Botulinum toxin type A is widely used for aesthetic treatment of mimic wrinkles. This study will investigate the safety and efficacy of NT 201 in the treatment of glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe glabellar frown lines at maximum frown ((severity score of 2 or 3 on Facial Wrinkle Scale(FWS)as assessed by the investigator's rating: 0 = 'none', 1 = 'mild', 2 = 'moderate', 3 = 'severe'
* Stable medical condition
* Age: between 18 and 65 years (inclusively)

Exclusion Criteria:

* Previous treatment with Botulinum toxin of any serotype in the upper third part of the face within the last 6 month
* Previous treatment with biodegradable fillers in the glabellar area within the last 12 month
* Previous insertion of permanent material in the glabellar area, including fat graft (regardless of the time between previous treatment and this study)
* Any surgery in the glabellar area including surgical removal of the corrugator, procerus, or depressor supercilii muscles or a combination of these, or scars in the glabellar area
* Any other planned cosmetic procedure in the upper third part of the face during the trial period
* Inability to substantially lessen glabellar frown lines even by physically spreading them apart
* Marked facial asymmetry or ptosis of eyelid and/or eyebrow
* History of facial nerve palsy
* Any infection in the area of the injection sites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Investigator's assessment | 4 weeks after initial injection session

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Imhof, MD, Principal Investigator — Ästhetische Dermatologie, Medico Palais Bad Soden
Locations (1):
- Dr. Matthias Imhof, Medico Palais Bad Soden, Bad Soden, Hesse, Germany

REFERENCES:
- [Result] Imhof M, Kuhne U. A Phase III Study of IncobotulinumtoxinA in the Treatment of Glabellar Frown Lines. J Clin Aesthet Dermatol. 2011 Oct;4(10):28-34. PMID 22010053